CLINICAL TRIAL: NCT06752759
Title: Nebulized Ketamine for the Treatment of Major Depressive Disorder in an Inpatient Setting: A Midazolam-controlled Randomized Controlled Trial
Brief Title: Nebulized Ketamine for the Treatment of Major Depressive Disorder in an Inpatient Setting
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Theresa Jacob, PhD, MPH (Other)
Responsible Party: Sponsor-Investigator, Theresa Jacob, PhD, MPH, Director of Research, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-06-05-MMC
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Severe Depression; Moderate Depression; Ketamine; Midazolam; Peripheral Nervous System Agents; Central Nervous System Agents; Neurotransmitter Agents; Physiologic Effects of Drugs; Sensory System Agents; Analgesics, Non-Narcotic; Anti-Inflammatory Agents, Non-Steroidal; Depressive Symptom; Hypnotics and Sedatives; Anti-anxiety Agents; Tranquilizing Agents; Psychotropic Drugs; Anesthetics Agent; GABA Modulators; GABA Agents
Keywords: Maimonides Medical Center; Psychiatry; Ketamine; Midazolam; Peripheral Nervous System Agents; Sensory System Agents; Anesthetics, Dissociative; Nebulized Medications for depression; GABA Agents
MeSH Terms: conditions — Depression | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nebulized Midazolam (Active Comparator): Midazolam used as active placebo. Dosage calculated by body weight at 0.03mg/kg
  Interventions: Drug: nebulized ketamine
- Nebulized Ketamine (Experimental): Ketamine dosage calculated by body weight at 1.5mg/kg
  Interventions: Drug: nebulized ketamine

INTERVENTIONS:
Drug: nebulized ketamine — The formulation of the study drug is administered via nebulizer in which the participants inhales the study drug. The dosage is calculated by body weight (1.5mg/kg).
  Other Names: Ketalar

SUMMARY:
This is a double blind active placebo controlled clinical trial for individuals within an inpatient setting with moderate to severe depression. The purpose of this study is to assess if nebulized ketamine can reduce depressive symptoms.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effect of ketamine formalized to be dispensed via inhalation, as an adjunct to concomitant medications and therapies on those with moderate to severe depression currently in an inpatient psychiatric unit. Investigators will examine the effects of nebulized ketamine on depressive symptoms.

This is a prospective double-blind placebo controlled study in which an active placebo, Midazolam, will be used. Participants will commit to either 4 visits or 5 visits depending on which treatment arm they are randomized into. All visits can be done remotely, however, days in which the participant will be dosed will have to be in person. During dosing days, the participant will be monitored for a minimum of two hours. Study participant's vitals will be collected at regular intervals during the observation period.

Adult psychiatry inpatients who are 18 years and older with a diagnosis of moderate to severe depression will be screened for enrollment by the study.

ELIGIBILITY:
Inclusion Criteria:

* All individuals 18 years and older within the Institution's inpatient Psychiatry Unit with a Montgomery-Asberg Depression Rating Scale score ≥ 20
* Must have a diagnosis of moderate to severe Major Depressive Disorder
* Structured Clinical Interview for DSM-5 (SCID-5) will be performed to confirm MDD diagnosis

Exclusion Criteria:

* Adult patients with an allergy to ketamine
* Adult patients with an allergy to Midazolam
* Individuals with a history of mania/hypomania or diagnosis of of bipolar disorder
* Patients on lithium and/or lamotrigine therapy
* Recent or current homicidal ideation with an intent to act
* MDD with psychotic features or current or past diagnosis of a psychotic disorder
* No substance use disorder in the preceding 3 months except nicotine or caffeine or a positive urine screen for substances (except cannabis)
* Diagnosis of obsessive-compulsive disorder, antisocial personality disorder, borderline personality disorder, posttraumatic stress disorder, intellectual disability, altered mental status, pregnant or breastfeeding patients,
* Patients on > 2 medications for hypertension
* Patients with uncontrolled hypertension (BP >140 mm Hg systolic and/or >90 mm Hg diastolic on two separate readings at the time of screening)
* Body weight of > 150kg
* Patients with history of congestive cardiac failure
* Day of presentation, patients with unstable vital signs (systolic blood pressure <90 or>160 mm Hg, pulse rate <50 or >150 beats/min, and respiration rate <10 or >30 breaths/min)
* Consumption of opioids within 24 hours of drug administration
* Acutely intoxicated patients will also be excluded

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms on the Montgomery-Åsberg Depression Rating Scale (MADRS) | 8-10 days
  Montgomery-Asberg Depression Rating Scale has a range from 0 to 60, where the lower score indicates the better health status. Change in mean total Montgomery Asberg Depression Rating Scale (MADRS) score from the baseline (pre-dose day 1 ), Day 2 and last day of assessments (Day 8 or Day 10)

SECONDARY OUTCOMES:
A change in depressive symptoms on the Montgomery-Åsberg Depression Rating Scale (MADRS) from the baseline (pre-dose on day 1) and 2 hours post-medication administration | 8-10 days
  Montgomery-Asberg Depression Rating Scale has a range from 0 to 60, where the lower score indicates the better health status. Change in mean total Montgomery-Asberg Depression Rating Scale prior to dose administration on Day 1, 2 hours after dose administration for each day.
Change in Beck Scale for Suicide Ideation | 24 hours
  Beck Scale for Suicide Ideation has a range from 0 to 42, where the lower score indicates the better health status. SSI score of ≥4, response which would be defined as SSI ≥50% below baseline - 2 hours post medication administration and remission defined as SSI score of ≥50% and lower than 4 - 24 hrs after medication administration of follow-up
Clinician-Administered Dissociative States Scale (CADSS) | 8-10 days
  Measurement of dissociative symptoms. Clinician Administered Dissociative States Scale (CADSS) comprises 23 subjective items, each on a 5 point scale, a "0" represents absence of any adverse events and "4" represents a severely bothersome side effect. A total score ranges from 0-92, a lower score indicates a better health status.
Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) | 8-10 days
  Overall side effects as measured by the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). SERSDA has 9 items, each graded on a five point scale, with "0" representing the absence of any adverse effects and "4" representing a severely bothersome side effect.
Maximal sedative effects using Modified Observer's Assessment of Alertness and Sedation ( MOAA/S) | 8-10 days
  Modified Observer's Alertness/Sedation Scale ( MOAA/S) uses a 6 point scale. A "0" indicates failure to respond to painful stimulus, "5" represents fully alert. .
Richmond Agitation-Sedation Scale (RASS) | 8-10 days
  Measurement of participant's consciousness with a rating ranging from +4 to -5. +4 represents "combative", +3 represents "Very agitated", +2 represents "Agitated" , +1 represents restless, 0 represents "Alert and calm", -1 represents "Drowsy", -2 represents "Light sedation", -3 represents "Moderate sedation", -4 represents "Deep sedation", and -5 represents "Unarousable".

CONTACTS AND LOCATIONS:
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Andrade C. Ketamine for Depression, 1: Clinical Summary of Issues Related to Efficacy, Adverse Effects, and Mechanism of Action. J Clin Psychiatry. 2017 Apr;78(4):e415-e419. doi: 10.4088/JCP.17f11567. PMID 28448702
- [Background] Dove D, Fassassi C, Davis A, Drapkin J, Butt M, Hossain R, Kabariti S, Likourezos A, Gohel A, Favale P, Silver M, Marshall J, Motov S. Comparison of Nebulized Ketamine at Three Different Dosing Regimens for Treating Painful Conditions in the Emergency Department: A Prospective, Randomized, Double-Blind Clinical Trial. Ann Emerg Med. 2021 Dec;78(6):779-787. doi: 10.1016/j.annemergmed.2021.04.031. Epub 2021 Jul 3. PMID 34226073
- [Background] Jonkman K, Dahan A, van de Donk T, Aarts L, Niesters M, van Velzen M. Ketamine for pain. F1000Res. 2017 Sep 20;6:F1000 Faculty Rev-1711. doi: 10.12688/f1000research.11372.1. eCollection 2017. PMID 28979762
- [Background] Wilkinson ST, Farmer C, Ballard ED, Mathew SJ, Grunebaum MF, Murrough JW, Sos P, Wang G, Gueorguieva R, Zarate CA Jr. Impact of midazolam vs. saline on effect size estimates in controlled trials of ketamine as a rapid-acting antidepressant. Neuropsychopharmacology. 2019 Jun;44(7):1233-1238. doi: 10.1038/s41386-019-0317-8. Epub 2019 Jan 17. PMID 30653192
- [Background] Drapkin J, Masoudi A, Butt M, Hossain R, Likourezos A, Motov S. Administration of Nebulized Ketamine for Managing Acute Pain in the Emergency Department: A Case Series. Clin Pract Cases Emerg Med. 2020 Jan 2;4(1):16-20. doi: 10.5811/cpcem.2019.10.44582. eCollection 2020 Feb. PMID 32064416
- [Background] Gao M, Rejaei D, Liu H. Ketamine use in current clinical practice. Acta Pharmacol Sin. 2016 Jul;37(7):865-72. doi: 10.1038/aps.2016.5. Epub 2016 Mar 28. PMID 27018176
- [Background] McIntyre RS, Rosenblat JD, Nemeroff CB, Sanacora G, Murrough JW, Berk M, Brietzke E, Dodd S, Gorwood P, Ho R, Iosifescu DV, Lopez Jaramillo C, Kasper S, Kratiuk K, Lee JG, Lee Y, Lui LMW, Mansur RB, Papakostas GI, Subramaniapillai M, Thase M, Vieta E, Young AH, Zarate CA Jr, Stahl S. Synthesizing the Evidence for Ketamine and Esketamine in Treatment-Resistant Depression: An International Expert Opinion on the Available Evidence and Implementation. Am J Psychiatry. 2021 May 1;178(5):383-399. doi: 10.1176/appi.ajp.2020.20081251. Epub 2021 Mar 17. PMID 33726522
- [Background] Yavi M, Lee H, Henter ID, Park LT, Zarate CA Jr. Ketamine treatment for depression: a review. Discov Ment Health. 2022;2(1):9. doi: 10.1007/s44192-022-00012-3. Epub 2022 Apr 15. PMID 35509843
- [Background] Kohtala S. Ketamine-50 years in use: from anesthesia to rapid antidepressant effects and neurobiological mechanisms. Pharmacol Rep. 2021 Apr;73(2):323-345. doi: 10.1007/s43440-021-00232-4. Epub 2021 Feb 20. PMID 33609274
- [Background] Park M, Niciu MJ, Zarate CA Jr. Novel Glutamatergic Treatments for Severe Mood Disorders. Curr Behav Neurosci Rep. 2015 Dec;2(4):198-208. doi: 10.1007/s40473-015-0050-5. Epub 2015 Oct 9. PMID 26824031
- [Background] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Background] Witkin JM, Martin AE, Golani LK, Xu NZ, Smith JL. Rapid-acting antidepressants. Adv Pharmacol. 2019;86:47-96. doi: 10.1016/bs.apha.2019.03.002. Epub 2019 Apr 24. PMID 31378256
- [Background] Henter ID, Park LT, Zarate CA Jr. Novel Glutamatergic Modulators for the Treatment of Mood Disorders: Current Status. CNS Drugs. 2021 May;35(5):527-543. doi: 10.1007/s40263-021-00816-x. Epub 2021 Apr 26. PMID 33904154
- [Background] Holma KM, Melartin TK, Haukka J, Holma IA, Sokero TP, Isometsa ET. Incidence and predictors of suicide attempts in DSM-IV major depressive disorder: a five-year prospective study. Am J Psychiatry. 2010 Jul;167(7):801-8. doi: 10.1176/appi.ajp.2010.09050627. Epub 2010 May 17. PMID 20478879
- [Background] Grunebaum MF, Galfalvy HC, Choo TH, Keilp JG, Moitra VK, Parris MS, Marver JE, Burke AK, Milak MS, Sublette ME, Oquendo MA, Mann JJ. Ketamine for Rapid Reduction of Suicidal Thoughts in Major Depression: A Midazolam-Controlled Randomized Clinical Trial. Am J Psychiatry. 2018 Apr 1;175(4):327-335. doi: 10.1176/appi.ajp.2017.17060647. Epub 2017 Dec 5. PMID 29202655
- [Background] Chung DT, Ryan CJ, Hadzi-Pavlovic D, Singh SP, Stanton C, Large MM. Suicide Rates After Discharge From Psychiatric Facilities: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2017 Jul 1;74(7):694-702. doi: 10.1001/jamapsychiatry.2017.1044. PMID 28564699
- [Background] Cavanagh JT, Carson AJ, Sharpe M, Lawrie SM. Psychological autopsy studies of suicide: a systematic review. Psychol Med. 2003 Apr;33(3):395-405. doi: 10.1017/s0033291702006943. PMID 12701661
- [Background] Pagan Colon IE, Kroin J, Kaushal S, Khan S, Alvarez Villalba CL. Increased Readmission Rates in Younger Male Patients Due to Suicidal Risk in Newly Diagnosed Depressive Disorders After Initiation of Serotonin Reuptake Inhibitors. Cureus. 2022 Nov 28;14(11):e31987. doi: 10.7759/cureus.31987. eCollection 2022 Nov. PMID 36589188
- [Background] Goodwin RD, Dierker LC, Wu M, Galea S, Hoven CW, Weinberger AH. Trends in U.S. Depression Prevalence From 2015 to 2020: The Widening Treatment Gap. Am J Prev Med. 2022 Nov;63(5):726-733. doi: 10.1016/j.amepre.2022.05.014. Epub 2022 Sep 19. PMID 36272761